CLINICAL TRIAL: NCT05590195
Title: Effect of PreforPro® (Prebiotic and Bacteriophage) on Urinary and Vaginal Health
Brief Title: Effect of PreforPro® on Urinary and Vaginal Health
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jeremy Burton (Other)
Collaborators: Deerland Enzymes (Industry); London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other); St. Joseph's Health Care London (Other)
Responsible Party: Sponsor-Investigator, Jeremy Burton, Principal Investigator, PhD, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BVPFB2021
Record Dates: First submitted 2022-10-06; First posted 2022-10-21 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Bacterial Vaginosis; Bacterial Infections; Bacterial Vaginosis | Vaginal | Microbiology; Vaginal Infection
MeSH Terms: conditions — Vaginosis, Bacterial; Bacterial Infections; Vaginitis

STUDY DESIGN:
Intervention Model Description: Double-blinded, randomized, placebo controlled study
Who Masked: Participant, Investigator
Masking Description: Neither participants nor study team will know which product the participants have been assigned. Unblinding can be requested from the pharmacy if necessary.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- PreforPro (Experimental): Preforpro Dosage form - capsule Dosage - participants will consume one capsule per day for 2 months treatment period
  Interventions: Drug: Preforpro
- Placebo (Placebo Comparator): placebo will come in a capsule, which has to be consumed one capsule per day for 2 months treatment period
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Preforpro — Preforpro will be investigated to improve vaginal health in women with BV.
  Arms: PreforPro
Other: Placebo — Placebo capsules manufactured to look like Preforpro capsules
  Other Names: Placebo for PreforPro
  Arms: Placebo

SUMMARY:
This study will investigate the effects of PreforPro® (prebiotic and bacteriophages (LH01-Myoviridae, LL5-Siphoviridae, T4D-Myoviridae, and LL12-Myoviridae, greater > 6.7 X 107 PFU/gram) on bacterial vaginosis.

DETAILED DESCRIPTION:
This is a double-blinded, placebo controlled study. Each study participant will be in the study for 90 days. During the first 28 days the participants will not take study product, and will collect samples for the study in order to act as their own controls. On day 29, participants will be randomized to intervention with either PreforPro® or placebo, which they will take once daily for the remaining 62 days. There will be a total of 5 study visits during which samples will be collected, a Quality of Life questionnaire will be completed at baseline and end of study visit.

Samples for the study are: vaginal swab, faecal sample, urine sample.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18-45 years old premenopausal (period within 6 months)
* Nugent score of 4-6 (intermediate) or 7-10 (BV)
* Have an ability to collect a clean urine sample
* Prescription and over the counter medication unchanged for > 30 days prior to the study. -Participants who are taking medications as needed (PRN) may be included if they began PRN usage >30 days prior to baseline
* Sexually active status of the participants can be either active or inactive
* Participants must agree to use a medically approved method of birth control (e.g. hormonal contraceptives, intrauterine devices, vasectomy/tubal ligation, barrier methods and double-barrier method) and must have negative pregnancy test results at screening and baseline

Exclusion Criteria:

* Faecal incontinence
* History of urinary fistula, bladder or kidney stones, interstitial cystitis, or cystoscopic abnormalities that could be malignant
* Neurogenic bladder
* A history of currently undergoing immunosuppressive drug therapy, chemotherapy, or radiation therapy
* Antibiotic and/or anti-fungal medication used within the last four weeks
* Oral probiotic supplement use within 2 weeks prior the study excluding yogurt
* Drug abuse
* Uncontrolled psychological disorders

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — This study is conducted in premenopausal females to improve the vaginal health in women with BV. Hence the participant eligibility is based on the gender.
Enrollment: 50 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
To change Nugent score in women with intermediate grade or BV | 3 months
  Vaginal swab is collected to determine the Nugent score, which is a The Nugent Score is a gram stain scoring system for vaginal swabs to diagnose bacterial vaginosis.
  Nugent scores between 7-10 is the standard diagnosis of BV and indicative of the absence of lactobacilli and a relative predominance of G. vaginalis and Mobiluncus spp. A Nugent score of 4-6 is indicative of intermediate BV. A Nugent score ≤ 3 means there is no BV.

SECONDARY OUTCOMES:
Determine whether the bacteriophage can translocate from the gastrointestinal system to genitourinary system. | 3 months
  Urine will be analyzed to determine the amount of antibiotic resistant genes by reverse transcriptase-quantitative polymerase chain reaction (qPCR). The Faecal sample will also be analyzed to determine bacteriophage counts by qPCR. These two tests will tell us if the bacteriophage was able to translocate between the two systems.
Determine if the microbiota in the gut and urinary system change | 3 months
  To determine this outcome the study team will test quantify and capture E. coli isolates from a urine sample. MSU microbiota analysis will be performed on the sample, and bacteriophage counts will be determined by qPCR.
Determine change in vaginal cell exfoliation. | 3 months
  Vaginal swab is collected to determine the amount of epithelial cell exfoliation.
Determine whether probiotics can translocate from the gastrointestinal system to genitourinary system. | 3 months
  MSU microbiota analysis will be performed on the urine and faecal sample to determine the species present in both samples.
Determine change in urogenital ATP levels. | 3 months
  Urine sample will be collected to quantify urogenital ATP level. A luminescent assay kit (BacTiter-Glo microbial cell viability assay; Promega, WI) will be used to quantify the amount of ATP. The Synergy H4 hybrid multimode microplate reader will be used to quantify the amount of ATP.

CONTACTS AND LOCATIONS:
Overall Officials: Jermy Burton, Principal Investigator — Lawson HRI